CLINICAL TRIAL: NCT03423537
Title: A Prospective, Multicenter, Double-blind, Placebo-controlled, Phase III Clinical Study, on the Efficacy and Safety of Low-dose hCG in a Short Protocol With GnRH Agonist and Ovarian Stimulation With Recombinant FSH (rFSH) During the Follicular Phase in Subfertile Women Undergoing ART
Brief Title: Low-dose HCG as an Adjunct to Ovarian Stimulation in Subfertile Women Undergoing ART
Acronym: HCG
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Inability for further recruitment, change of position of the principal investigator, COVID-19 pandemic
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, Siristatidis Charalampos, MD, PhD, Associate Professor in Obstetrics and Gynecology, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: hCG-GR-001-2016; 2016-005208-24 (EudraCT Number)
Record Dates: First submitted 2018-01-21; First posted 2018-02-06 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2020-09

CONDITIONS: HCG; IVF; Pregnancy Rates; ART; Chorionic Gonadotropin
MeSH Terms: interventions — Chorionic Gonadotropin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 [HCG (+) group] (Experimental): "Group 1" will indicate the application of the protocol by adding hCG with the initiation of standard GnRH agonist protocol for IVF / ICSI with rFSH
  Interventions: Drug: hCG
- Group 2 [placebo] (Placebo Comparator): "Group 2" will indicate the application of the standard GnRH agonist protocol without the addition of hCG, but placebo, instead
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: hCG — the addition of hCG (Pregnyl®, MSD Greece) will begin with the administration of gonadotrophin at a dose of 100 IU per day, administered subcutaneously, and will continue until the administration of hCG for follicular maturation.
  Other Names: Pregnyl
  Arms: Group 1 [HCG (+) group]
Drug: Placebo — 100IU per day containing N/S 0.9% will be injected
  Arms: Group 2 [placebo]

SUMMARY:
The objective of this prospective randomized clinical trial is to investigate whether the addition of low-dose hCG to a short GnRH-agonist protocol for IVF and ovarian stimulation with rFSH from the onset of the follicular phase and throughout stimulation in sub fertile women undergoing IVF, improves pregnancy rates.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized, double-blind, placebo-controlled, two parallel group of patients, Phase IIIb clinical study to test the efficacy and safety of adding low-dose hCGs in a short protocol with GnRH agonist and ovarian stimulation with recombinant FSH (rFSH) from the onset of the follicular phase and throughout the duration of stimulation in enrolled women to the increase in the rate of clinical pregnancies.

Main end point will be the rate of clinical pregnancy (positive heart rate at 7 weeks of gestation in the ultrasound), while secondary endpoints will be

* The number of follicles (> 11,> 14,> 18 mm) on the day of triggering with hCG
* The thickness of the endometrium on the day of follicular maturation
* Live birth rates
* Automatic abortion rates (loss of pregnancy after positive heart function up to 20 weeks of gestation)
* The rate of ongoing pregnancy (positive heart function after 12 weeks of gestation),
* The percentage of ovarian hyperstimulation syndrome (after triggering) with hCG for the next 2 weeks
* The rate of multiple pregnancy.

Participants will be randomly divided into two groups: the intervention group (Group 1) and the control group (Group 2). Randomization will be done using sealed envelopes marked "Group 1" and "Group 2". The randomization list will be prepared centrally for the four participating clinics (research centers) and there will be a "stratification" per center, per 30, respectively, and will be shared among the participants.

"Group 1" will indicate the application of the protocol by adding hCG with the initiation of controlled ovarian stimulation protocol for IVF / ICSI with rFSH, and "Group 2" will indicate the application of the conventional protocol without the addition of hCG .

Each patient's assignment to a treatment group will be made by calling the unit's midwife who will have 2 envelopes with the above indications and who will not be present when the pair is informed by 2 members of the research team.

ELIGIBILITY:
Inclusion Criteria:

1. Age: between 35 and 40 years of age,
2. Physiological menstrual cycles (24-35 day cycle),
3. Normal endocrine function (normal PRL and TSH, FSH ≤ 15 IU / ml),
4. Transvaginal ultrasound (TVS) without pathological findings,
5. Free personal medical history,
6. Indication for IVF / ICSI (NICE, 2016)
7. 1st or 2nd IVF / ICSI cycle

Exclusion Criteria:

1. Endocrine or metabolic disorders, e.g. PCO (S)
2. Pathology of the uterus and / or endometrium,
3. Pelvic inflammatory disease (PID),
4. Basal FSH levels> 15 IU / ml,
5. Surgery in the ovaries,
6. Body Mass Index (BMI) ≥ 35 kg / m2,
7. Age: <35 years &> 41 years old

Ages: 35 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
number of transferred embryos | 21 days after the beginning of ovarian stimulation
  number of high quality transferred embryos at day 3
The rate of clinical pregnancy | 7 weeks after the initiation of treatment
  Positive heart rate at 7 weeks of gestation in ultrasound

SECONDARY OUTCOMES:
Number of follicles | 2 weeks after the initiation of treatment
  (> 11,> 14,> 18 mm) on the day of triggering with hCG
The thickness of the endometrium | 2 weeks after the initiation of treatment
  On the day of follicular maturation (triggering) with hCG
Automatic abortion rates - miscarriage | up to 20 weeks of gestation
  (Lss of pregnancy after positive heart function up to 20 weeks of gestation
The percentage of ovarian hyperstimulation syndrome | 2 weeks after the hCG triggering
  After triggering with hCG

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Siristatidis, Ass Prof, Principal Investigator — National and Kapodistrian University of Athens
Locations (1):
- 3rd Department of Obstetrics and Gynecology, Assisted Reproduction Unit, Athens, Chaidari, Greece

REFERENCES:
- [Result] Drakakis P, Loutradis D, Beloukas A, Sypsa V, Anastasiadou V, Kalofolias G, Arabatzi H, Kiapekou E, Stefanidis K, Paraskevis D, Makrigiannakis A, Hatzakis A, Antsaklis A. Early hCG addition to rFSH for ovarian stimulation in IVF provides better results and the cDNA copies of the hCG receptor may be an indicator of successful stimulation. Reprod Biol Endocrinol. 2009 Oct 13;7:110. doi: 10.1186/1477-7827-7-110. PMID 19825188
- [Result] Gomaa H, Casper RF, Esfandiari N, Chang P, Bentov Y. Addition of low dose hCG to rFSh benefits older women during ovarian stimulation for IVF. Reprod Biol Endocrinol. 2012 Aug 6;10:55. doi: 10.1186/1477-7827-10-55. PMID 22866896
- [Result] Martins WP, Vieira AD, Figueiredo JB, Nastri CO. FSH replaced by low-dose hCG in the late follicular phase versus continued FSH for assisted reproductive techniques. Cochrane Database Syst Rev. 2013 Mar 28;2013(3):CD010042. doi: 10.1002/14651858.CD010042.pub2. PMID 23543584
- [Result] Beretsos P, Partsinevelos GA, Arabatzi E, Drakakis P, Mavrogianni D, Anagnostou E, Stefanidis K, Antsaklis A, Loutradis D. "hCG priming" effect in controlled ovarian stimulation through a long protocol. Reprod Biol Endocrinol. 2009 Aug 31;7:91. doi: 10.1186/1477-7827-7-91. PMID 19719843
- See also: Current guidelines — https://www.nice.org.uk/guidance/cg156